CLINICAL TRIAL: NCT06912386
Title: A Randomized Two-Way Crossover Comparison Study of Pain Relief From Dysmenorrhea Employing taVNS and Sham Stimulation
Brief Title: Pain Relief From Dysmenorrhea Employing taVNS
Acronym: taVNS-DYSM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Electronic Science and Technology of China (Other)
Responsible Party: Principal Investigator, stefania, Prof. Stefania Ferraro, University of Electronic Science and Technology of China
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: UESTC-neuSCAN-99; taVNS_DYSM_01 (Other: UESTC)
Record Dates: First submitted 2025-03-24; First posted 2025-04-04 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-03

CONDITIONS: Dysmenorrhea Primary
Keywords: Dysmenorrhea; transauricular vagal nerve stimulation; Pain
MeSH Terms: conditions — Dysmenorrhea; Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- taVNS - transauricular vagal nerve stimulation (Experimental): Transauricular Vagus Nerve Stimulation (taVNS) will be applied in the tragus with the following parameters:
  Pulse width: 500 microseconds; Frequency: 25 Hz; Stimulation cycle: 30 seconds on, 30 seconds off; Duration: 15 minutes per session; Current: Adjustable between 0 and 10 mA, with step increments of 0.1 mA.
  Interventions: Device: taVNS
- SHAM stimulation (Sham Comparator): Stimulation of the earlobe will be applied with the following parameters:
  Pulse width: 500 microseconds; Frequency: 25 Hz; Stimulation cycle: 30 seconds on, 30 seconds off; Duration: 15 minutes per session; Current: Adjustable between 0 and 10 mA, with step increments of 0.1 mA.
  Interventions: Device: SHAM stimulation

INTERVENTIONS:
Device: taVNS — Intervention Name: Transauricular Vagus Nerve Stimulation (taVNS)
  Intervention Description:
  Participants will receive transauricular vagus nerve stimulation on the tragus. Frequency: 2 sessions per day (one at 10 AM and one at 6 PM). Duration: Each session will last 15 minutes. Treatment Cycle: Stimulation will be applied for 5 days each month, starting 2 days before the expected beginning of the menstrual cycle, for a total of 2 months. The participants will adjust the level of maximum stimulation they considered painless.
  Arms: taVNS - transauricular vagal nerve stimulation
Device: SHAM stimulation — Intervention Name: SHAM stimulation of the earlobe. Participants will receive SHAM stimulation on the earlobe, which does not stimulate the vagus nerve.
  Frequency: 2 sessions per day (one at 10 AM and one at 6 PM). Duration: Each session will last 15 minutes. Treatment Cycle: Placebo stimulation will be applied for 5 days each month, starting 2 days before the expected beginning of the menstrual cycle, for a total of 2 months. The participants will adjust the level of maximum stimulation they considered painless.
  Arms: SHAM stimulation

SUMMARY:
The goal of this clinical trial is to determine if transauricular vagal nerve stimulation (taVNS) is effective in treating moderate dysmenorrhea. The main question it aims to answer is:

• Does taVNS reduce the number of times participants suffering from dysmenorrhea need to use rescue medication during menstruation? Researchers will compare taVNS stimulation with a sham stimulation (a look-alike procedure that does not stimulate the vagus nerve) to assess whether taVNS is effective in treating moderate dysmenorrhea.

Participants will:

* Undergo taVNS for 2 months and sham stimulation for another 2 months, each for 5 days per month, starting 2 days before the expected beginning of their menstrual cycle.
* Visit the clinic twice a month for checkups and tests.
* Keep a diary to record their pain levels and the number of times they use rescue medication.
* Undergo functional magnetic resonance imagine two times (one after the end of the first use of taVNS and another after the end of the first use of SHAM stimulation).

ELIGIBILITY:
Inclusion Criteria:

* Regular menstrual cycle (28 days ± 7 days);
* Average moderate menstrual pain (with 4 - 7 NRS scores);
* History of over-the-counter (OTC) analgesic use for the treatment of menstrual pain (at least 1 IBUPROFEN for the first two days);
* 4 consecutive monthly menstrual cycles;
* Non-pregnant status;
* Agrees to use adequate birth control during the trial;
* Otherwise, healthy;
* Agree not to participate in any other clinical trial while enrolled in this trial ;
* No facial or ear pain, no recent ear trauma, no metal implants including pacemakers;
* Normal ECG, Heart Rate and Blood Pressure (systolic BP 105-130, diastolic BP 60-90, heart rate per min at rest 60-85);

Exclusion Criteria:

* Currently under medications (except for analgesic medication for menstrual cycle);
* Use of oral contraceptive;
* Secondary cause for dysmenorrhea (i.e., endometriosis, adenomyosis, uterine fibroids, or infection);
* Unstable or serious illness (e.g., kidney, liver, GIT, heart conditions, diabetes, thyroid gland function, lung conditions, chronic asthma, diagnosed psychological or mood disorder, hypertension, any bleeding disorders, recent surgery, or concurrent blood thinning treatment);
* Current malignancy or treatment for malignancy within the previous 2 years;
* Pregnant or lactating women;
* Active smokers, nicotine use, or drug (prescription or illegal substances) abuse;
* Chronic past and/or current alcohol use (>14 alcoholic drinks per week);
* Any condition that in the opinion of the investigator, makes the participant unsuitable for inclusion;
* Unwilling or unable to comply with protocol;
* Active genitourinary infection in the last four weeks;
* Unable to read or comprehend the informed consent;
* Unwilling to complete study procedures;
* Participated in any other clinical trial during the past 1 month;
* Personal or family history of seizure, mood, or cardiovascular disorders;
* Allergic reaction to surface electrodes.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 20 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Reduction the use of rescue medications | During the first 3 days of menstrual
  Significative reduction in the number of cases of rescue medication after the treatment employing the taVNS in respect to the sham condition.

SECONDARY OUTCOMES:
Reduction in acute and mean menstrual pain severity | During the first 3 days of menstrual
  Significative reduction in acute and mean (across the 3 days) menstrual pain severity assessed via Numeric Rating Scale (NRS) after the treatment employing the taVNS in respect to the sham condition.
Reduction in menstrual pain severity at the Short form McGill Pain Questionnarie | During the first 3 days of menstrual
  Reduction in menstrual pain severity employing using the Short form McGill pain questionnaire during the experimental condition in comparison to the sham condition
Changes in affective symptoms | First day of stimulation, last day of stimulation.
  Decrease of the score in at least one if the following scale: in Trait Anxiety Inventory (STAI), Beck's Depression Inventory II, Positive and Negative Affect Schedule (PANAS) and Pain Catastrophizing Scale (PCS).
Changes in fMRI signal in the mesocorticolimbic system | After the first month application of the taVNS and of the SHAM stimulation
  Changes in fMRI signal in the areas of the mesocorticolimibic system during the execution of a reward fMRI task (Monetary incentive delay task, Kuntson et al., 2001).

CONTACTS AND LOCATIONS:
Locations (1):
- UESTC, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Yes
Primary and secondary outcomes
Supporting Information: Study Protocol
Time Frame: IPD will be available at the end of the relevant analyses with not limit of time.
Access Criteria: IPD will be available on the platform OSF